CLINICAL TRIAL: NCT04820413
Title: Faecal Microbiota Transplantation Using Stool From Normal Pouch Function Donor in the Treatment of Chronic Pouchitis
Brief Title: Faecal Microbiota Transplantation From Normal Pouch Function Donor in the Treatment of Chronic Pouchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery (Other)
Responsible Party: Sponsor-Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, Professor of surgery, Consultant surgeon, DMSc, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MicroPouch-NP
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Pouchitis; Inflammatory Bowel Diseases; Ulcerative Colitis
Keywords: FMT; Microbiota
MeSH Terms: conditions — Pouchitis; Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT (Experimental)
  Interventions: Other: Faecal microbiota transplantation

INTERVENTIONS:
Other: Faecal microbiota transplantation — FMT by daily enema with donor faeces

SUMMARY:
Patients with chronic pouchitis is disabled by bloody diarrhoea and abdominal pain often followed by fever. Pouchitis is an inflammation in a pouch, a reservoir formed by the small intestine in the management of the chronic inflammatory bowel disease, ulcerative colitis. The standard treatment for pouchitis is intensive broad-spectrum antibiotics for a longer period. However, the treatment often fails after repeated treatments. Studies show that patients with pouchitis have an altered composition of the gut microbiota compared to healthy individuals and patients with a pouch without inflammation. As shown by several studies, faecal microbiota transplantation (FMT) with administration of faeces from healthy donors can alter the microbiota. Treatment with faecal microbiota transplantation to chronic pouchitis has been investigated in several clinical trials with mixed results. It is however still uncertain if faecal microbiota transplantation using stool from healthy individuals with a colon is optimal, or if stool from patient with a normally functioning pouch should be used.

The study primary aims to investigate if transplantation of faeces from patient with a normal pouch function can induce clinical remission in patients with chronic pouchitis.

DETAILED DESCRIPTION:
Hypothesis:

Gut dysbiosis plays a significant causal role in chronic pouchitis. Modulating the gut microbiota using FMT with stool from a normal function pouch patient has a clinical effect by inducing clinical remission in patients with chronic pouchitis.

Objective of the study:

The aim of the trial is to investigate if transplantation (FMT) of faeces from a patient with a normally functioning pouch can induce clinical remission in patients with chronic pouchitis.

Study design:

The project is designed as a single-center, open-label, treatment study.

Methods:

Faecal microbiota transplantation is performed with faeces from a donor with a normally functioning pouch. Potential donors are recruited from the Department of Gastrointestinal Surgery, Aalborg University Hospital, Denmark. They are screened for a various of infectious diseases by serum analysis (haematology, inflammation, liver and kidney function, HIV, Hepatitis, Cytomegalovirus, Epstein Barr virus and HbA1c) and faeces analysis (calprotectin, Clostridium difficile (PCR), enteric pathogenic bacteria and antibiotic-resistant bacteria, parasites, cysts, and viruses). Furthermore, the potential donors will complete an extensive questionnaire regarding general health, risk factors and medical history, before they can be included as faecal donors in the project. The screening procedure is based on recommendation from the European FMT Working Group.

The transplantation is performed by enemas, which contain faeces from the faecal donor.

Initial before the treatment with FMT, the patient will be invited for serum analysis (CRP, leukocytes) and faecal analysis (calprotectin, C.difficile, enteric pathogenic bacteria), followed by a pouchoscopy with collection of biopsies. Materials from serum- and faecal analysis and biopsies will be stored for later analysis purpose. The patient will further complete questionnaires concerning symptoms and quality of life. The stage of disease will be evaluated based on the acknowledged questionnaire for pouchitis called Pouchitis Disease Activity Index (PDAI) score.

The treatment begins after all the initial examinations, and the patient will be treated during one month. The treatment consists of daily enema infusion, which contain faeces from the faecal donor. During the treatment, the patient will daily record symptoms related to pouchitis (diarrhea, abdominal pain, bleeding per rectum, fever, general discomfort) and possible adverse effects to the treatment.

At the end of treatment, the patient will meet to a follow-up examination including serum analysis (CRP, leukocytes) and faecal analysis (calprotectin), pouchoscopy incl. biopsies, and the questionnaires applied before the treatment. Materials from serum- and faecal analysis and biopsies will be stored for later analysis.

The patient will be followed up after additional 1,3, 6 and 12 months to evaluate the long term effect of the transplantation. The consumption of antibiotics during the first year will be recorded. In case of lacking effect of faecal microbiota transplantation, the patient is offered standard antibiotic treatment for pouchitis, and will leave the study.

Faecal samples and biopsies collected in the study will be analyzed for the composition of the microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with a J-pouch
* PDAI ≥ 7
* Established diagnosis of chronic pouchitis (≥3 times of pouchitis within the last year, symptoms more than 4 weeks despite antibiotic treatment)
* Antibiotic treatment for pouchitis (ciprofloxacin and/or metronidazole) within the 3 months

Exclusion Criteria:

* Immunosuppression
* Pregnancy or breastfeeding
* Evidence of intestinal pathogen bacteria in the stool at inclusion visit
* Any severe or newly diagnosed concomitant cardiovascular, hepatic, intestinal, renal, endocrine, pulmonary, dental disease with inflammation or psychiatric disorder, which, in the opinion of the investigator, might have an influence on the patient's compliance or the interpretation of the results
* Probiotic intake within the last 2 weeks prior to study intervention
* Participation in another clinical trial within the previous 30 days before baseline
* Serious food allergies with earlier anaphylactic reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving clinical remission assessed by PDAI | 4 weeks
  Clinical remission is defined as PDAI<7

SECONDARY OUTCOMES:
Number of patients achieving clinical response assessed by PDAI | 4 weeks
  Clinical response is defined as reduction of PDAI score >2
Engraftment of the donor microbiota in the patients | 4 weeks
  Assessed by beta-diversity

CONTACTS AND LOCATIONS:
Overall Officials: Ole Thorlacius-Ussing, Professor, Study Chair — Aalborg University Hospital
Locations (1):
- Department of Gastrointestinal Surgery, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No